CLINICAL TRIAL: NCT05570344
Title: Repetitive Transcranial Magnetic Stimulation With and Without Text4Support for the Treatment of Resistant Depression: Patient-centered Multicentral Randomized Controlled Pilot Trial. Protocol.
Brief Title: rTMS With and Without Text4Support for the Treatment of Resistant Depression.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00122696
Record Dates: First submitted 2022-09-19; First posted 2022-10-06 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Depressive Disorder, Treatment-Resistant
Keywords: Repetitive Transcranial Magnetic Stimulation; Treatment of Resistant Depression; Patient - Centered Randomized Controlled Pilot Trial; Supportive Text messages (Text4Support)
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: This is a prospective, Multicenter, two-arm randomized controlled trial. 200 patients diagnosed with resistant depression in psychiatric care clinics in Edmonton, Alberta, and Nova Scotia, Canada will be randomized to one of two conditions: (1) enrolment in rTMS sessions alone (2) enrolment in the rTMS sessions plus Text4Support.
Who Masked: Outcomes Assessor
Masking Description: Because it will not be possible for participants to be blinded, treatment allocation will be made explicit to them as soon as randomization is concluded. Primary outcome assessors will be blinded to treatment group allocation by not involving them in discussions about study participants and not granting them access to the database which contains the randomization code. After data collection is complete, all data will undergo a blind review for the purposes of finalizing the planned analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enrolment in rTMS sessions alone (Active Comparator): All study participants will be scheduled to receive 30 sessions of rTMS treatment for 6 weeks as pre-established by the Alberta Health Services Strategic Clinical Network for Addiction and Mental Health and Nova Scotia Health.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- Enrolment in rTMS sessions plus Text4Support (Experimental): Participants in the rTMS plus Text4Support group of the study would be assisted by a study team member assigned that purpose to register onto the Text4Support program. The process would require all participants to input their phone numbers into the Text4Support platform that will be used to deliver the daily messages. Starting a day after enrollment, participants will receive daily supportive text messages designed by mental health therapists, clinical psychologists, psychiatrists, and mental health service users. These messages are based on cognitive behavior therapy principles crafted to enhance positively the mood of its users with depressive symptoms and other related mental health problems of concern. The messages will be pre-programmed into a software program that will deliver the messages to participants automatically to the participants' mobile phones at 10 AM (Mountain Time) and 12 PM (Atlantic Time), and each participant will receive these messages continuously for 6 weeks.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS) Plus Text4Support

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — rTMS uses powerful (1.0-2.5 Tesla), focused magnetic field pulses to induce electrical currents in neural tissue noninvasively, via an inductor coil placed against the scalp.
  Arms: Enrolment in rTMS sessions alone
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) Plus Text4Support — rTMS uses powerful (1.0-2.5 Tesla), focused magnetic field pulses to induce electrical currents in neural tissue noninvasively, via an inductor coil placed against the scalp.
  Text4Support:
  Text4Support is one of the ResilienceNHope suites of supportive text messaging programs delivered by the Global Psychological eHealth Foundation [80]. The program allows users to receive daily supportive text messages which have been written by a team of cognitive-behavioral therapists and mental health professionals in collaboration with users of mental health services. The aim of this Text4Support depression program is to enhance positively the mood of patients with clinical depression. The program operates through the use of positive reinforcement to correct distorted or negative thought patterns.
  Arms: Enrolment in rTMS sessions plus Text4Support

SUMMARY:
This study is a multicenter prospective, parallel design, two-arm, rater-blinded randomized controlled pilot trial. Participants will be randomly assigned to one of two treatment conditions. In the first condition, treatment consists of rTMS sessions combined with Text4Support. The second condition is made up of the treatment as usual (rTMS sessions alone). The recruitment process is scheduled to last 12 months. It will involve active treatment for six weeks and follow-up period observation periods of 1,3, and 6 months for participants in both arms of the study. Participants will be recruited from four different centers for this project. Two centers (the Addiction and Mental Health clinic and the Alberta day hospital) will be from the large, sociodemographic diverse city of Edmonton in Alberta Western Canada. The remaining two centers will be in Halifax and Annapolis Valley in Nova Scotia, Canada.

DETAILED DESCRIPTION:
Objective: This study aims to assess the initial comparative clinical effectiveness of rTMS with and without the Text4Support program as an innovative patient-centered intervention for the management of participants diagnosed with TRD.

Methods: This study is a multicentered prospective, parallel-design, two-arm, rater-blinded randomized controlled pilot trial. The recruitment process is scheduled to last 12 months. It will involve active treatment for six weeks, observation, and a follow-up period of six months for participants in both arms of the study. In total, 200 participants diagnosed with TRD at rTMS care clinics in Edmonton, Alberta, and rTMS clinics in Halifax, Nova Scotia will be randomized to one of two treatment arms (rTMS sessions alone and rTMS sessions plus Text4Support intervention. Participants in each group will be made to complete evaluation measures at baseline, one month, three months, and six months. The primary outcome measure will be the mean change to scores on the Patient Health Questionnaire (PHQ-9). Patient service utilization data and clinician-rated measures will also be used to gauge patient progress. Patient data will be analyzed with descriptive statistics, repeated measures, and correlational analyses.

Interventions: Study participants will be randomized to one of the treatment interventions (rTMS alone or rTMS plus Text4Support). During the introductory visit to the study sites, participants in both arms of the study will be given a detailed orientation about the rTMS application, and all procedures and activities within each visit will be explained to them. As part of their participation in the rTMS program, all patients will be made to complete some standard measures. Participants will be invited to the various rTMS clinics a week before the commencement of the rTMS sessions to enable them to undergo motor threshold (MT) assessments. The MT assessment is essential in that it aids in the selection of the required stimulation intensity for each patient for inclusion in the treatment. MT assessment is a measure of the minimum intensity of TMS output needed to elicit a motor response in the participating TRD patients in at least 50% of all attempts.

The MT assessments will be conducted by the rTMS team of experts within the rTMS clinics in the various treatment centers and may consist of psychiatrists, nurses, and other healthcare professionals with the requisite knowledge to do so. Each TMS assessment session will take about 3-5 minutes, and the total time will be within 35-45 minutes. This visit timeline will be the same for all study participants. Overall, all study participants will be scheduled to receive 30 sessions of rTMS treatment for 6 weeks as pre-established by the Alberta Health Services Strategic Clinical Network for Addiction and Mental Health and Nova Scotia Health.

Additionally, participants in the rTMS plus Text4Support group of the study will be assisted by a study team member assigned that purpose to register on to the Text4Support program. The process will require all participants in this arm of the study to input their phone numbers into the Text4Support platform that will be used to deliver the daily messages. Starting a day after enrollment, participants will receive daily supportive text messages designed by mental health therapists, clinical psychologists, psychiatrists, and mental health service users. These messages are based on cognitive behavior therapy principles crafted to enhance positively the mood of its users with depressive symptoms and other related mental health problems of concern. The messages will be pre-programmed into a software program that will deliver the messages to participants automatically to the participants' mobile phones at 10 AM (Mountain Time) and 12 PM (Atlantic Time), and each participant will receive these messages continuously for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 and above and diagnosed with MDD based upon the criteria of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) and who have at least failed two or more standard antidepressant treatments during the current episode. Participants may be on psychotropic medications including antidepressants, antipsychotics, benzodiazepines, and anticonvulsants. They must have a good understanding of the English language. Must have access to a smartphone and be able to receive and read text messages. Must be willing to provide written informed consent upon acceptance into the study.

Exclusion Criteria:

* Patients below the age of 18.
* Having diagnosis such as the following conditions (current unless otherwise stated): A neurological disorder, including a history of seizures, having primary or secondary tumors in the central nervous system, cerebrovascular disease, stroke, cerebral aneurysm, movement disorder,
* Having a current psychotic disorder such as substance-induced psychosis, psychotic disorder due to a medical condition, or MDD with psychotic features at the time of screening
* Having a current personality disorder that may hinder the patient's participation in this research or may have the potential of affecting cognition and ability to fully participate in the study.
* Having a learning disability as per identified through medical history or by the investigator during the assessment process.
* Participants involved in any drug or device clinical trial within the last six weeks before the screening visit and/or involvement in another clinical trial for the duration of this study.
* Pregnant and breastfeeding women.
* Identification and/or the sudden appearance of any condition or instance from the mentioned above and based on the expertise of the investigators that have the potential to hinder the progress and completion and/or become a confounding factor on the outcome assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
The Patient Health Questionnaire (PHQ-9) | Baseline
  With 9 items, the PHQ-9 is half the length of many other depression measures, has comparable sensitivity and specificity, and it's made up of the actual 9 criteria upon which the diagnosis of depressive disorders according to the DSM-IV is based. This instrument has the potential to establish major depressive disorder diagnoses as well as grading the severity of depressive symptom
The Patient Health Questionnaire (PHQ-9) | 1 month
  With 9 items, the PHQ-9 is half the length of many other depression measures, has comparable sensitivity and specificity, and it's made up of the actual 9 criteria upon which the diagnosis of depressive disorders according to the DSM-IV is based. This instrument has the potential to establish major depressive disorder diagnoses as well as grading the severity of depressive symptom
The Patient Health Questionnaire (PHQ-9) | 3 months
  With 9 items, the PHQ-9 is half the length of many other depression measures, has comparable sensitivity and specificity, and it's made up of the actual 9 criteria upon which the diagnosis of depressive disorders according to the DSM-IV is based. This instrument has the potential to establish major depressive disorder diagnoses as well as grading the severity of depressive symptom
The Patient Health Questionnaire (PHQ-9) | 6 months
  With 9 items, the PHQ-9 is half the length of many other depression measures, has comparable sensitivity and specificity, and it's made up of the actual 9 criteria upon which the diagnosis of depressive disorders according to the DSM-IV is based. This instrument has the potential to establish major depressive disorder diagnoses as well as grading the severity of depressive symptom

SECONDARY OUTCOMES:
Generalized Anxiety Disorders Scale (GAD-7) | Baseline
  The GAD-7 scale is calculated by assigning scores of 0, 1, 2, and 3 to the response categories, respectively, of "not at all," "several days," "more than half the days," and "nearly every day." GAD-7 total score for the seven items ranges from 0 to 21. (0-4: minimal anxiety, 5-9: mild anxiety, 10-14: moderate anxiety, and 15-21: severe anxiety)
Generalized Anxiety Disorders Scale (GAD-7) | 1 month
  The GAD-7 scale is calculated by assigning scores of 0, 1, 2, and 3 to the response categories, respectively, of "not at all," "several days," "more than half the days," and "nearly every day." GAD-7 total score for the seven items ranges from 0 to 21. (0-4: minimal anxiety, 5-9: mild anxiety, 10-14: moderate anxiety, and 15-21: severe anxiety)
Generalized Anxiety Disorders Scale (GAD-7) | 3 months
  The GAD-7 scale is calculated by assigning scores of 0, 1, 2, and 3 to the response categories, respectively, of "not at all," "several days," "more than half the days," and "nearly every day." GAD-7 total score for the seven items ranges from 0 to 21. (0-4: minimal anxiety, 5-9: mild anxiety, 10-14: moderate anxiety, and 15-21: severe anxiety)
Generalized Anxiety Disorders Scale (GAD-7) | 6 months
  The GAD-7 scale is calculated by assigning scores of 0, 1, 2, and 3 to the response categories, respectively, of "not at all," "several days," "more than half the days," and "nearly every day." GAD-7 total score for the seven items ranges from 0 to 21. (0-4: minimal anxiety, 5-9: mild anxiety, 10-14: moderate anxiety, and 15-21: severe anxiety)
Columbia Suicide Severity Rating Scale | Baseline
  To assess suicidal ideation as symptom variable. Suicidal Ideation Score: The maximum suicidal ideation category (1-5 on the C- SSRS) present at the assessment. Assign a score of 0 if no ideation is present.
Columbia Suicide Severity Rating Scale | 1 month
  To assess suicidal ideation as symptom variable. Suicidal Ideation Score: The maximum suicidal ideation category (1-5 on the C- SSRS) present at the assessment. Assign a score of 0 if no ideation is present.
Columbia Suicide Severity Rating Scale | 3 months
  To assess suicidal ideation as symptom variable. Suicidal Ideation Score: The maximum suicidal ideation category (1-5 on the C- SSRS) present at the assessment. Assign a score of 0 if no ideation is present.
Columbia Suicide Severity Rating Scale | 6 months
  To assess suicidal ideation as symptom variable. Suicidal Ideation Score: The maximum suicidal ideation category (1-5 on the C- SSRS) present at the assessment. Assign a score of 0 if no ideation is present.
The World Health Organization - Five Well-Being Index (WHO-5) | Baseline
  To assess the mental wellbeing as a functional variable. The total raw score, ranging from 0 to 25, is multiplied by 4 to give the final score, with 0 representing the worst imaginable well-being and 100 representing the best imaginable well-being.
The World Health Organization - Five Well-Being Index (WHO-5) | 1 month
  To assess the mental wellbeing as a functional variable. The total raw score, ranging from 0 to 25, is multiplied by 4 to give the final score, with 0 representing the worst imaginable well-being and 100 representing the best imaginable well-being.
The World Health Organization - Five Well-Being Index (WHO-5) | 3 months
  To assess the mental wellbeing as a functional variable. The total raw score, ranging from 0 to 25, is multiplied by 4 to give the final score, with 0 representing the worst imaginable well-being and 100 representing the best imaginable well-being.
The World Health Organization - Five Well-Being Index (WHO-5) | 6 months
  To assess the mental wellbeing as a functional variable. The total raw score, ranging from 0 to 25, is multiplied by 4 to give the final score, with 0 representing the worst imaginable well-being and 100 representing the best imaginable well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Agyapong, MD, Ph.D, Principal Investigator — Division of Community Psychiatry, University of Alberta
Locations (2):
- Canada (2):
  - Edmonton Mental Health Clinic, Edmonton, Alberta
  - Nova Scotia Health - Abbie J. Lane Memorial Building QEII Health Sciences Centre, Halifax, Nova Scotia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agyapong VIO, Juhas M, Ohinmaa A, Omeje J, Mrklas K, Suen VYM, Dursun SM, Greenshaw AJ. Randomized controlled pilot trial of supportive text messages for patients with depression. BMC Psychiatry. 2017 Aug 2;17(1):286. doi: 10.1186/s12888-017-1448-2. PMID 28768493
- [Background] Agyapong VI, Milnes J, McLoughlin DM, Farren CK. Perception of patients with alcohol use disorder and comorbid depression about the usefulness of supportive text messages. Technol Health Care. 2013;21(1):31-9. doi: 10.3233/THC-120707. PMID 23358057
- [Background] Agyapong VI, Mrklas K, Juhas M, Omeje J, Ohinmaa A, Dursun SM, Greenshaw AJ. Cross-sectional survey evaluating Text4Mood: mobile health program to reduce psychological treatment gap in mental healthcare in Alberta through daily supportive text messages. BMC Psychiatry. 2016 Nov 8;16(1):378. doi: 10.1186/s12888-016-1104-2. PMID 27821096
- [Background] Rush AJ, Trivedi MH, Ibrahim HM, Carmody TJ, Arnow B, Klein DN, Markowitz JC, Ninan PT, Kornstein S, Manber R, Thase ME, Kocsis JH, Keller MB. The 16-Item Quick Inventory of Depressive Symptomatology (QIDS), clinician rating (QIDS-C), and self-report (QIDS-SR): a psychometric evaluation in patients with chronic major depression. Biol Psychiatry. 2003 Sep 1;54(5):573-83. doi: 10.1016/s0006-3223(02)01866-8. PMID 12946886
- [Background] Tanner JA, Hensel J, Davies PE, Brown LC, Dechairo BM, Mulsant BH. Economic Burden of Depression and Associated Resource Use in Manitoba, Canada. Can J Psychiatry. 2020 May;65(5):338-346. doi: 10.1177/0706743719895342. Epub 2019 Dec 13. PMID 31835904